CLINICAL TRIAL: NCT06419777
Title: Strict Versus Permissive Threshold for Initiation of Pharmacotherapy in Gestational Diabetes Mellitus (GDM) With Glucometer Use - A Randomized Control Trial (START1)
Brief Title: Strict Versus Permissive Thresholds for Initiation of Pharmacotherapy in Gestational Diabetes
Acronym: START 1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iRISID-2024-2999
Record Dates: First submitted 2024-05-09; First posted 2024-05-17 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Gestational Diabetes; Pregnancy Related
Keywords: gestational diabetes; pregnancy; insulin; Initiation of medication
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance | interventions — Insulin; Insulin Glargine; Insulin Lispro; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strict Arm (Active Comparator): The strict threshold is defined as two abnormal values or more over a one-week period (two fasting values elevated, two of the same post prandial values elevated, or 1 fasting and 1 post prandial value elevated)
  Interventions: Drug: Insulin
- Permissive (Active Comparator): The permissive threshold is defined as 50% of values elevated over 1 week (50% of overall fasting values, 50% of postprandial values, or 50% of overall values).
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin will be used in gestational diabetics to control blood glucose levels
  Other Names: Lantus; Lispro; NPH; Levemir; Humalog

SUMMARY:
The aim of our study is to compare neonatal and maternal outcomes using different thresholds for the initiation and titration of pharmacotherapy for gestational diabetes (GDM). Our goal is to compare a strict and permissive threshold. The strict threshold is defined as two abnormal values or more over a one-week period (two fasting values elevated, two of the same post prandial values elevated, or 1 fasting and 1 post prandial value elevated), whereas the permissive threshold is defined as 50% of values elevated over 1 week (50% of overall fasting values, 50% of postprandial values, or 50% of overall values).

DETAILED DESCRIPTION:
Pregnancy is a state of insulin resistance to ensure that the growing fetus has ample nutrition. Gestational Diabetes (GDM) develops in pregnant patients with pancreatic dysfunction that leads to impairment of glucose tolerance.

Various studies have examined the benefit of treatment for GDM, including the 2005 Australian Carbohydrate Intolerance Study in Pregnant Women (ACHOIS) and the 2009 Landon et al randomized controlled trials. These studies found that treatment was associated with a significant reduction in newborn complications of perinatal death, shoulder dystocia, large for gestational age infants, cesarean delivery, and birth trauma. The specific threshold value for initiation and up-titration of medical therapy is unknown. Lack of evidence leads to a wide variation in clinical practice of pharmacological initiation and titration for GDM. A systematic review and meta-analysis by Caissutti in 2019 analyzed criteria for initiating pharmacotherapy for GDM and noted the following: 12 of 15 trials initiated pharmacotherapy after 1-2 abnormal values over 1-2 weeks, 2 studies initiated pharmacotherapy after 50% of overall values were abnormal, and 1 study initiated pharmacotherapy after 30% of overall values were abnormal. However, there have been no randomized controlled trials of head-to-head comparison of different thresholds.

The aim of our study is to compare neonatal and maternal outcomes using different thresholds for the initiation and titration of pharmacotherapy for gestational diabetes. Our goal is to compare a strict and relaxed threshold. The strict threshold is defined as two abnormal values or more over a one week period (two fasting values elevated, two of the same post prandial values elevated, or 1 fasting and 1 post prandial value elevated), whereas the relaxed threshold is defined as 50% of values elevated over 1 week (50% of overall fasting values, 50% of postprandial values, or 50% of overall values).

ELIGIBILITY:
Inclusion Criteria:

* Live, non-anomalous fetus
* Literacy in English, Spanish, Mandarin, or Arabic
* Patients are also required to provide consent, demonstrate an understanding of the purpose of the study, and agree to the study protocol.

Exclusion Criteria:

* <18 years at EDD
* pre-existing diabetes or diagnosis of GDM before 24 weeks
* multi-fetal gestation
* known major fetal anomaly
* known allergy to insulin
* chronic maternal corticosteroid use
* diagnosis of GDM based on finger sticks alone
* patients who have contraindication to oral glucose tolerance test
* a primary language other than English, Spanish, Mandarin, or Arabic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Neonatal Composite Outcome | First 28 days of birth
  neonatal composite including the following measures: large for gestational age (LGA) of neonate defined as birth weight >90th percentile for gestational age using the Fenton growth chart, hypoglycemia o defined as glucose <40 mg/dL <48 hours after birth or glucose, hyperbilirubinemia, stillbirth or neonatal death, birth trauma

SECONDARY OUTCOMES:
Neonatal Outcome: Gestational Age of Birth | Delivery Time
  Gestational age at delivery in weeks and days
Neonatal Outcome: APGAR Score | At 1 minute of life and at 5 min of life
  Scoring system provided a standardized assessment for infants after delivery from 0-10
Neonatal Outcome: Birthweight | Delivery Time
  Birthweight in grams, Macrosomia (birthweight >4000g, Small for gestational age (<10th percentile based on Fenton Growth Charts)
Neonatal Outcome: Brachial Plexus Injury | Delivery Time
  Brachial plexus nerves in neonate are torn, stretched, or compressed at delivery
Neonatal Outcome: Respiratory distress | Within first 24 hours after delivery
  Breathing difficulties after birth requiring supplemental oxygen, mask, intubation, and/or surfactant
Neonatal Outcome: Admission to Neonatal intensive Care Unit | From delivery to discharge from NICU
  Admission to neonatal intensive care unit (NICU)
Maternal Outcomes: Maternal hypoglycemia | Initiation of insulin to delivery
  Maternal episode of hypoglycemia < 60 mg/dL throughout the pregnancy
Maternal Outcomes: Shoulder Dystocia | At Delivery
  An obstetric emergency where the anterior fetal shoulder becomes stuck on the maternal pubic symphysis, delaying the birth of the baby's body.
Maternal Outcomes: Obstetric anal sphincter injury (OASIS) | At Delivery
  3rd degree and 4th degree perineal injuries
Maternal Outcomes: Operative Delivery | At Delivery
  Vacuum-assisted and Forcep-assisted vaginal Delivery
Maternal Outcomes: Cesarean Delivery | At Delivery
  Cesarean birth
Maternal Outcomes: Postpartum hemorrhage | Within 24 hours of delivery
  Defined as cumulative blood loss ≥1000 mL, or bleeding associated with signs/symptoms of hypovolemia within 24 hours of the birth process
Maternal Outcomes: Hypertensive Disorders of Pregnancy | From gestational age of 20 weeks during pregnancy to 6 weeks postpartum
  Hypertensive disorders of pregnancy: gestational hypertension, Preeclampsia without severe features, Pre-eclampsia with severe features, severe range blood pressures defined as (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥110 mmHg), symptoms of central nervous dysfunction, thrombocytopenia with Platelet count <100,000 platelets/microL, hepatic abnormalities, kidney impairment, and or pulmonary edema

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Rochester Medical Center, Rochester, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kunarathnam V, Vadakekut ES, Mahdy H. Gestational Diabetes. 2025 Sep 15. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK545196/ PMID 31424780
- [Result] Catalano PM, Hauguel-De Mouzon S. Is it time to revisit the Pedersen hypothesis in the face of the obesity epidemic? Am J Obstet Gynecol. 2011 Jun;204(6):479-87. doi: 10.1016/j.ajog.2010.11.039. Epub 2011 Feb 2. PMID 21288502
- [Result] Gregory EC, Ely DM. Trends and Characteristics in Gestational Diabetes: United States, 2016-2020. Natl Vital Stat Rep. 2022 Jul;71(3):1-15. PMID 35877134
- [Result] Metzger BE, Persson B, Lowe LP, Dyer AR, Cruickshank JK, Deerochanawong C, Halliday HL, Hennis AJ, Liley H, Ng PC, Coustan DR, Hadden DR, Hod M, Oats JJ, Trimble ER; HAPO Study Cooperative Research Group. Hyperglycemia and adverse pregnancy outcome study: neonatal glycemia. Pediatrics. 2010 Dec;126(6):e1545-52. doi: 10.1542/peds.2009-2257. Epub 2010 Nov 15. PMID 21078733
- [Result] ACOG Practice Bulletin No. 190: Gestational Diabetes Mellitus. Obstet Gynecol. 2018 Feb;131(2):e49-e64. doi: 10.1097/AOG.0000000000002501. PMID 29370047
- [Result] Crowther CA, Hiller JE, Moss JR, McPhee AJ, Jeffries WS, Robinson JS; Australian Carbohydrate Intolerance Study in Pregnant Women (ACHOIS) Trial Group. Effect of treatment of gestational diabetes mellitus on pregnancy outcomes. N Engl J Med. 2005 Jun 16;352(24):2477-86. doi: 10.1056/NEJMoa042973. Epub 2005 Jun 12. PMID 15951574
- [Result] Landon MB, Spong CY, Thom E, Carpenter MW, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Lain KY, Sorokin Y, Peaceman AM, Tolosa JE, Anderson GB; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. A multicenter, randomized trial of treatment for mild gestational diabetes. N Engl J Med. 2009 Oct 1;361(14):1339-48. doi: 10.1056/NEJMoa0902430. PMID 19797280
- [Result] Hartling L, Dryden DM, Guthrie A, Muise M, Vandermeer B, Donovan L. Benefits and harms of treating gestational diabetes mellitus: a systematic review and meta-analysis for the U.S. Preventive Services Task Force and the National Institutes of Health Office of Medical Applications of Research. Ann Intern Med. 2013 Jul 16;159(2):123-9. doi: 10.7326/0003-4819-159-2-201307160-00661. PMID 23712381
- [Result] Davitt C, Flynn KE, Harrison RK, Pan A, Palatnik A. Current practices in gestational diabetes mellitus diagnosis and management in the United States: survey of maternal-fetal medicine specialists. Am J Obstet Gynecol. 2021 Aug;225(2):203-204. doi: 10.1016/j.ajog.2021.04.263. Epub 2021 May 14. No abstract available. PMID 34000260
- [Result] Caissutti C, Saccone G, Ciardulli A, Berghella V. Very tight vs. tight control: what should be the criteria for pharmacologic therapy dose adjustment in diabetes in pregnancy? Evidence from randomized controlled trials. Acta Obstet Gynecol Scand. 2018 Mar;97(3):235-247. doi: 10.1111/aogs.13257. Epub 2017 Dec 14. PMID 29125636
- [Result] Harrison RK, Cruz M, Wong A, Davitt C, Palatnik A. The timing of initiation of pharmacotherapy for women with gestational diabetes mellitus. BMC Pregnancy Childbirth. 2020 Dec 11;20(1):773. doi: 10.1186/s12884-020-03449-y. PMID 33308193
- [Result] Landy HJ, Gomez-Marin O, O'Sullivan MJ. Diagnosing gestational diabetes mellitus: use of a glucose screen without administering the glucose tolerance test. Obstet Gynecol. 1996 Mar;87(3):395-400. doi: 10.1016/0029-7844(95)00460-2. PMID 8598962
- [Result] Harper LM, Mele L, Landon MB, Carpenter MW, Ramin SM, Reddy UM, Casey B, Wapner RJ, Varner MW, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Caritis SN, Sorokin Y, Peaceman AM, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Carpenter-Coustan Compared With National Diabetes Data Group Criteria for Diagnosing Gestational Diabetes. Obstet Gynecol. 2016 May;127(5):893-898. doi: 10.1097/AOG.0000000000001383. PMID 27054932
- [Result] Blum AK. Insulin Use in Pregnancy: An Update. Diabetes Spectr. 2016 May;29(2):92-7. doi: 10.2337/diaspect.29.2.92. PMID 27182178
- [Result] Fenton TR, Kim JH. A systematic review and meta-analysis to revise the Fenton growth chart for preterm infants. BMC Pediatr. 2013 Apr 20;13:59. doi: 10.1186/1471-2431-13-59. PMID 23601190